CLINICAL TRIAL: NCT07080996
Title: Effect of Biofeedback Tongue Strengthening Program on Tongue Pressure and Swallowing Performance in Elderly With Abnormal Tongue Pressure
Brief Title: Effect of Biofeedback Tongue Strengthening Program on Tongue Pressure and Swallowing Performance
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Surachart Thongchoomsin, Lecturer, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MU-CIRB 2025/037.2201
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Presbyphagia; Abnormal Tongue Pressure
Keywords: Elderly; Presbyphagia; Dysphagia; Tongue Pressure; Biofeedback
MeSH Terms: conditions — Deglutition Disorders | interventions — Biofeedback, Psychology; Endurance Training

STUDY DESIGN:
Intervention Model Description: All participants are randomly assigned to either the strengthening training or endurance training group using a computer.
Who Masked: Participant, Outcomes Assessor
Masking Description: This research is a double-blind study, in which both participants and the assessor are blinded to the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strengthening training group (Experimental): Participants trained their tongue strength three times a week for four weeks.
  Interventions: Combination Product: Strengthening training with biofeedback
- Endurance training group (Active Comparator): Participants trained their tongue endurance three times a week for four weeks.
  Interventions: Combination Product: Endurance training with biofeedback

INTERVENTIONS:
Combination Product: Strengthening training with biofeedback — Participants in this group trained their tongue strength with the Iowa Oral Performance Instrument (IOPI), completing 3 sets of 10 repetitions at 80% of their maximum.
  Arms: Strengthening training group
Combination Product: Endurance training with biofeedback — Participants in this group trained their tongue endurance with the Iowa Oral Performance Instrument (IOPI), completing 3 sets of 20 repetitions at 60% of their maximum.
  Arms: Endurance training group

SUMMARY:
Aging is often accompanied by a decline in bodily functions, including the swallowing process. Tongue-strengthening exercises have been shown to improve tongue strength and thickness in healthy adults and the elderly, thereby supporting swallowing function. Consistent exercise is key to preventing muscle weakness and preserving their ability to swallow. However, there is limited research on the effects of tongue-strengthening exercises that explores varying intensities and repetitions in elderly with impaired tongue pressure. Consequently, the objective of this study is to investigate the effect of biofeedback tongue strengthening program on tongue pressure and swallowing performance in elderly with abnormal tongue pressure. The results will serve as valuable data for selecting effective interventions to improve tongue strength and swallowing.

DETAILED DESCRIPTION:
Sample size calculation: A sample size of 52 participants was determined for this study, accounting for a 20% dropout rate. The calculation was performed using G*Power software (version 3.1.7), based on an effect size of 0.87. This value was derived from a previous study by Van den Steen et al. (21), which measured the difference in mean tongue pressure strength between training and control groups. With an effect size of 0.87, considered a large effect, a minimum of 44 participants was required to achieve 80% statistical power at a significance level of 0.05. Statistical analysis: IBM SPSS Statistics will be used for all data analysis. A chi-squared test and Mann-Whitney U test will be performed to compare the baseline characteristics of participants between the two groups. A two-way ANOVA will be used to analyze differences between the two groups (strengthening training and endurance training) across the three time points (Baseline, Post-test after one day, and Post-test after one month). Subsequently, a Wilcoxon signed-rank test will be used to identify significant changes within each group at each time point.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or older.
* No cognitive impairment, as screened by the Mini-Mental State Examination (MMSE) with a score of 24 or higher.
* Elderly with abnormal tongue pressure have an anterior maximum isometric tongue pressure (MIP) average of less than 30 kilopascals.

Exclusion Criteria:

* Diagnosed with head and neck cancers, a neurological disorder, or other conditions that affect the tongue muscle strength and training.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-02-24 (Estimated); Study Completion 2026-03-24 (Estimated)

PRIMARY OUTCOMES:
Tongue pressure | Baseline, Post-test after one day of training, Post-test after one month of training
  The Iowa Oral Performance Instrument (IOPI Medical LCC, Redmond, WA USA) was used to measure maximum anterior and posterior tongue pressure, as well as tongue pressure during swallowing.
Eating Assessment Tool-10 (EAT-10) score | Baseline, Post-test after one day of training, Post-test after one month of training
  The EAT-10 is used to assess swallowing difficulties. The 10 items are scored from 0 to 4, with higher scores indicating more severe dysphagia.
Functional Oral Intake Scale (FOIS) | Baseline, Post-test after one day of training, Post-test after one month of training
  The FOIS is a 7-point ordinal scale describing the functional level of oral intake of food and liquids.
Mann Assessment of Swallowing Ability (MASA) score | Baseline, Post-test after one day of training, Post-test after one month of training
  The MASA is a standardized clinical swallowing examination, specifically developed as a diagnostic test for the presence of oropharyngeal dysphagia. The total score of the MASA is 200 points and the cutoff value is 177 points. The results of the MASA are interpreted as no abnormality (≥178), mild dysphagia (168-177), moderate dysphagia (139-167), and severe dysphagia (≤138).
Water swallowing test | Baseline, Post-test after one day of training, Post-test after one month of training
  The Water Swallow Test is a clinical instrument designed to assess swallowing function. A participant is seated and provided with a cup containing 150 mL of water at a standard temperature. The total time required to ingest the liquid is then recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
We will share IPD when we receive the consent from participants.

REFERENCES:
- [Background] Nakao Y, Yamashita T, Honda K, Katsuura T, Hama Y, Nakamura Y, Ando K, Ishikura R, Kodama N, Uchiyama Y, Domen K. Association Among Age-Related Tongue Muscle Abnormality, Tongue Pressure, and Presbyphagia: A 3D MRI Study. Dysphagia. 2021 Jun;36(3):483-491. doi: 10.1007/s00455-020-10165-4. Epub 2020 Aug 2. PMID 32743742
- [Background] Delfraissy JF. [New therapeutic strategies in HIV infection]. Presse Med. 1997 Apr 19;26(13):612-4. No abstract available. French. PMID 9180874
- [Background] Thomas SH, Stone CK, Bryan-Berge D, Hunt RC. Effect of an in-flight helicopter environment on the performance of ALS interventions. Air Med J. 1994 Jan;13(1):9-12. doi: 10.1016/S1067-991X(05)80004-5. PMID 10131003
- [Background] Stenke L, Reizenstein P, Lindgren JA. Leukotrienes and lipoxins--new potential performers in the regulation of human myelopoiesis. Leuk Res. 1994 Oct;18(10):727-32. doi: 10.1016/0145-2126(94)90053-1. PMID 7934130
- [Background] Thiels E, Kanterewicz BI, Knapp LT, Barrionuevo G, Klann E. Protein phosphatase-mediated regulation of protein kinase C during long-term depression in the adult hippocampus in vivo. J Neurosci. 2000 Oct 1;20(19):7199-207. doi: 10.1523/JNEUROSCI.20-19-07199.2000. PMID 11007876
- [Background] State HIV-positive physician policy. N J Med. 1993 Feb;90(2):91. No abstract available. PMID 8464581
- [Background] Kiehl MG, Ostermann H, Meyer J, Kienast J. Nitric oxide synthase inhibition by L-NAME in leukocytopenic patients with severe septic shock. Intensive Care Med. 1997 May;23(5):561-6. doi: 10.1007/s001340050373. PMID 9201529
- [Background] White MS. On the scene: University of Cincinnati Hospital. The disease of chemical dependency: recovery to restoration. Nurs Adm Q. 1985 Winter;9(2):38-41. No abstract available. PMID 3844107
- [Background] Sylvest-Hansen B. [WHO's global AIDS program]. Sjukskoterskan. 1989 Spring:4-6. No abstract available. Swedish. PMID 2749282
- [Background] Arcaroli J, Kupfner J, Yum HK, Shenkar R, Park JS, Abraham E. Lipopolysaccharide-induced neutrophil gene expression under in vivo or in vitro conditions. Chest. 2002 Mar;121(3 Suppl):76S. doi: 10.1378/chest.121.3_suppl.76s. No abstract available. PMID 11893694
- [Background] Reed TJ, Allen HS Jr. Supreme Court relaxes exclusive contract rules in antitrust decision. Trustee. 1984 Jun;37(6):34-8. PMID 10266797
- [Background] Hirel B, Chesne C, Pailheret JP, Guillouzo A. Expression of differentiation markers in human adult keratinocytes cultured in submerged conditions. In Vitro Cell Dev Biol Anim. 1994 Jun;30A(6):372-8. doi: 10.1007/BF02634357. PMID 7522100
- [Background] Tamminga CA, Conley RR. The application of neuroimaging techniques to drug development. J Clin Psychiatry. 1997;58 Suppl 10:3-6. PMID 9265909
- [Background] Keith CG, Doyle LW. Retinopathy of prematurity in extremely low birth weight infants. Pediatrics. 1995 Jan;95(1):42-5. PMID 7770307
- [Background] Yamazaki M, Maebayashi Y, Miyaki K. The isolation of secalonic acid A from Aspergillus ochraceus cultured on rice. Chem Pharm Bull (Tokyo). 1971 Jan;19(1):199-201. doi: 10.1248/cpb.19.199. No abstract available. PMID 5544365
- [Background] Smaoui S, Langridge A, Steele CM. The Effect of Lingual Resistance Training Interventions on Adult Swallow Function: A Systematic Review. Dysphagia. 2020 Oct;35(5):745-761. doi: 10.1007/s00455-019-10066-1. Epub 2019 Oct 14. PMID 31612288
- [Background] Satake A, Kobayashi W, Tamura Y, Oyama T, Fukuta H, Inui A, Sawada K, Ihara K, Noguchi T, Murashita K, Nakaji S. Effects of oral environment on frailty: particular relevance of tongue pressure. Clin Interv Aging. 2019 Sep 12;14:1643-1648. doi: 10.2147/CIA.S212980. eCollection 2019. PMID 31564844
- [Background] Imamura Y, Chebib N, Ohta M, Maria Schulte-Eickhoff R, Mekki M, Schimmel M, Arakawa I, Graf C, Sato Y, Muller F. Validation of a novel diagnostic tool for decreased tongue pressure. J Oral Rehabil. 2021 Nov;48(11):1219-1225. doi: 10.1111/joor.13232. Epub 2021 Sep 12. PMID 34425018
- [Background] Hughes TA, Wiles CM. Clinical measurement of swallowing in health and in neurogenic dysphagia. QJM. 1996 Feb;89(2):109-16. doi: 10.1093/qjmed/89.2.109. PMID 8729551
- [Background] Ohira M, Ishida R, Maki Y, Ohkubo M, Sugiyama T, Sakayori T, Sato T. Evaluation of a dysphagia screening system based on the Mann Assessment of Swallowing Ability for use in dependent older adults. Geriatr Gerontol Int. 2017 Apr;17(4):561-567. doi: 10.1111/ggi.12755. Epub 2016 May 16. PMID 27195778
- [Background] Shimizu A, Fujishima I, Maeda K, Wakabayashi H, Nishioka S, Ohno T, Nomoto A, Shigematsu T, Kayashita J; Japanese Working Group on Sarcopenic Dysphagia. Effect of low tongue pressure on nutritional status and improvement of swallowing function in sarcopenic dysphagia. Nutrition. 2021 Oct;90:111295. doi: 10.1016/j.nut.2021.111295. Epub 2021 Apr 28. PMID 34107332
- [Background] Szynkiewicz SH, Kamarunas E, Drulia T, Nobriga CV, Griffin L, O'Donoghue CR. A Randomized Controlled Trial Comparing Physical and Mental Lingual Exercise for Healthy Older Adults. Dysphagia. 2021 Jun;36(3):474-482. doi: 10.1007/s00455-020-10164-5. Epub 2020 Aug 8. PMID 32770381
- [Background] Yano J, Yamamoto-Shimizu S, Yokoyama T, Kumakura I, Hanayama K, Tsubahara A. Effects of anterior tongue strengthening exercises on posterior tongue strength in healthy young adults. Arch Oral Biol. 2019 Feb;98:238-242. doi: 10.1016/j.archoralbio.2018.11.028. Epub 2018 Nov 28. PMID 30522043
- [Background] Burkhead LM, Sapienza CM, Rosenbek JC. Strength-training exercise in dysphagia rehabilitation: principles, procedures, and directions for future research. Dysphagia. 2007 Jul;22(3):251-65. doi: 10.1007/s00455-006-9074-z. Epub 2007 Apr 25. PMID 17457549
- [Background] Van den Steen L, Vanderwegen J, Guns C, Elen R, De Bodt M, Van Nuffelen G. Tongue-Strengthening Exercises in Healthy Older Adults: Does Exercise Load Matter? A Randomized Controlled Trial. Dysphagia. 2019 Jun;34(3):315-324. doi: 10.1007/s00455-018-9940-5. Epub 2018 Sep 12. PMID 30209561
- [Background] Waldon EG, Broadhurst E. Construct validity and reliability of the Music Attentiveness Screening Assessment (MASA). J Music Ther. 2014 Summer;51(2):154-70. doi: 10.1093/jmt/thu008. Epub 2014 Jun 27. PMID 25013945
- [Background] Belafsky PC, Mouadeb DA, Rees CJ, Pryor JC, Postma GN, Allen J, Leonard RJ. Validity and reliability of the Eating Assessment Tool (EAT-10). Ann Otol Rhinol Laryngol. 2008 Dec;117(12):919-24. doi: 10.1177/000348940811701210. PMID 19140539
- [Background] Kunieda K, Ohno T, Fujishima I, Hojo K, Morita T. Reliability and validity of a tool to measure the severity of dysphagia: the Food Intake LEVEL Scale. J Pain Symptom Manage. 2013 Aug;46(2):201-6. doi: 10.1016/j.jpainsymman.2012.07.020. Epub 2012 Nov 15. PMID 23159683
- [Background] Tanaka T, Takahashi K, Hirano H, Kikutani T, Watanabe Y, Ohara Y, Furuya H, Tetsuo T, Akishita M, Iijima K. Oral Frailty as a Risk Factor for Physical Frailty and Mortality in Community-Dwelling Elderly. J Gerontol A Biol Sci Med Sci. 2018 Nov 10;73(12):1661-1667. doi: 10.1093/gerona/glx225. PMID 29161342
- [Background] Robbins J, Levine R, Wood J, Roecker EB, Luschei E. Age effects on lingual pressure generation as a risk factor for dysphagia. J Gerontol A Biol Sci Med Sci. 1995 Sep;50(5):M257-62. doi: 10.1093/gerona/50a.5.m257. PMID 7671027
- [Background] Nicosia MA, Hind JA, Roecker EB, Carnes M, Doyle J, Dengel GA, Robbins J. Age effects on the temporal evolution of isometric and swallowing pressure. J Gerontol A Biol Sci Med Sci. 2000 Nov;55(11):M634-40. doi: 10.1093/gerona/55.11.m634. PMID 11078092
- [Background] Aoki Y, Kabuto S, Ozeki Y, Tanaka T, Ota K. The effect of tongue pressure strengthening exercise for dysphagic patients. Jpn J Compr Rehabil Sci. 2015;6:129-136.
- [Background] Hara K, Tohara H, Kobayashi K, Yamaguchi K, Yoshimi K, Nakane A, Minakuchi S. Age-related declines in the swallowing muscle strength of men and women aged 20-89 years: A cross-sectional study on tongue pressure and jaw-opening force in 980 subjects. Arch Gerontol Geriatr. 2018 Sep-Oct;78:64-70. doi: 10.1016/j.archger.2018.05.015. Epub 2018 May 31. PMID 29902686
- [Background] Robbins J, Hamilton JW, Lof GL, Kempster GB. Oropharyngeal swallowing in normal adults of different ages. Gastroenterology. 1992 Sep;103(3):823-9. doi: 10.1016/0016-5085(92)90013-o. PMID 1499933
- [Background] Ortega O, Martin A, Clave P. Diagnosis and Management of Oropharyngeal Dysphagia Among Older Persons, State of the Art. J Am Med Dir Assoc. 2017 Jul 1;18(7):576-582. doi: 10.1016/j.jamda.2017.02.015. Epub 2017 Apr 12. PMID 28412164